CLINICAL TRIAL: NCT05222217
Title: Gatekeeper™ Prostheses Implants for Patients With Gas Incontinence and Soiling
Brief Title: Gatekeeper for Soiling and Gas Incontinence
Status: Completed | Type: Observational
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Principal Investigator, Arantxa Muñoz-Duyos, Clinical Chief of General and Digestive Surgery, Hospital Mutua de Terrassa
Other Study IDs: P21/0001
Record Dates: First submitted 2021-12-24; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Gas Incontinence; Soilings, Fecal
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Device: Gatekeeper — Six polyacrylonitrile prostheses (THD Gatekeeper™ Delivery System, THD SpA, Correggio, Italy) were implanted under 3D-EUS control through a 5mm perianal incision at 1, 3, 5, 7, 9 and 11 o'clock in lithotomy position, and located in the upper-middle intersphincteric space of the anal canal, using a specifically designed system.

SUMMARY:
Faecal incontinence has a broad spectrum of symptoms. Some patients only suffer commonly considered mild symptoms: gas incontinence and soiling, but patients' quality of life is significantly impaired. Although several treatments for faecal incontinence are available, this subgroup of patients are difficult to treat, and no therapeutic alternative has been clearly defined.

The aim of this study is to evaluate Gatekeeper™ treatment for this subgroup of patients with faecal incontinence, not studied before.

Consecutive case series single-centre study. Patients with mainly soiling and/or gas incontinence were treated with polyacrylonitrile prostheses

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years old
* with at least 6 months of GI and/or soiling
* non-responding to conservative treatment and biofeedback.

Exclusion Criteria:

* complete solid and liquid FI
* common Bristol score > 4
* malignant diseases
* chronic diarrhoea
* inflammatory bowel disease
* acute anorectal disease
* rectal prolapse
* neurological disease,
* obstructive defecation syndrome
* low anterior resection syndrome,
* previous pelvic radiation,
* any anaesthetic contraindication
* St. Mark's score > 12
* external anal sphincter lesion > 30º.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients' selection was based on clinical history, physical examination, preoperative 3D-endoanal ultrasound (EUS) and a continence diary recorded for 21 days. Patients with previous history of chronic diarrhoea were evaluated by the gastroenterology team and if needed, fibre supplementation or other medical treatment was used to obtain a Bristol score of 3-4 before entering the study
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in the number of gas incontinence and soiling episodes | 6, 12 and 24 months after surgery
  Each patient completes a three-week continence diary specifically recording gas incontinence and soiling episodes at baseline and before every follow-up visit.
Changes in incontinence symptoms | 6, 12 and 24 months after surgery
  Evaluation of incontinence symptoms with the St. Mark's Incontinence Score.
  Score from 0 to 24, where 0 means "complete continence" and 24 means "severe fecal incontinence"
Patient's Subjective Perception | 6, 12 and 24 months after surgery
  Changes in patient subjective evaluation using a Visual Analogue Scale (VAS).
  Score from 0 to 10, where 0 means "no problem" and 10 means "severe problem and alteration of my quality of life"

SECONDARY OUTCOMES:
Changes in prostheses location | baseline and one month after surgery
  Prostheses migration was defined as displacement of the prosthesis to the suprasphincteric space detected during the follow-up, detected with 3D-Endoanal Ultrasound.
Differences in anal pressures | baseline and three months after surgery
  Measurement of differences in anal testing pressures using a four-channel manometer

IPD SHARING:
Plan to Share IPD: No